CLINICAL TRIAL: NCT07306819
Title: Flexible Ureteroscopy Using a Tip-Bendable Suction Ureteral Access Sheath Versus Mini-Percutaneous Nephrolithotomy for the Treatment of 2-3 cm Renal Stones: A Randomized Controlled Trial
Brief Title: Comparison Between Two Methods for Renal Stone Treatment Mini Percutaneous Nephrolithotomy and Flexible Ureteroscopy With Suction Sheath
Acronym: mini-PCNL/FANS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed M Hasab Allah, resident of urology, Ahmed Maher Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MS 725/2025
Record Dates: First submitted 2025-11-28; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-11

CONDITIONS: Stone;Renal; Stone, Urinary; Stone, Kidney; Stone Clearance
MeSH Terms: conditions — Nephrolithiasis; Urinary Calculi; Kidney Calculi

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mini-PCNL (Experimental): Under general anesthesia, a 6 Fr ureteral catheter will be placed into the target ureter via cystoscopy, and bladder drainage will be achieved with a 16 Fr Foley catheter. The patient will then be repositioned to the prone position. Percutaneous renal access will be obtained by puncturing the selected calyx with an 18-gauge coaxial needle under fluoroscopic or ultrasound guidance. Tract dilation will be performed using fascial dilators up to 20 Fr then the mini-PCNL sheath (mini-Amplatz sheath) will be inserted and the mini nephroscope 12 to 15 Fr will be used. If multiple nephrostomy tracts are required for stone removal, the same approach will be repeated for each tract. Stone fragmentation will be carried out with a pneumatic lithotripter.
  At the end of the procedure, a 6 Fr double-J ureteral stent will be inserted for 4 weeks, and whether to place a nephrostomy tube will be determined at the discretion of the operating surgeon.
  Interventions: Procedure: mini-percutaneous nephrolithotomy
- FURS with Tip-Bendable Suction Sheath (Experimental): under general anesthesia with the patient in the lithotomy position. A 6 Fr ureteral catheter will first be placed into the ureter, followed by retrograde pyelography to assess the upper urinary tract. A guidewire will then be advanced into the renal pelvis. either a 12/14 Fr or 11/13 Fr tip-bendable S-UAS will be inserted. If insertion is not possible due to ureteral narrowing, a smaller 10/12 Fr UAS will be attempted. if failed, a double-J stent will be placed and the procedure terminated, with a second session scheduled 4 weeks later. fURS will be performed using digital flexible ureteroscopes either 8.5 Fr or 7.5 Fr according to UAS size; an 8.5-Fr scope for a 12/14 Fr UAS, and a 7.5-Fr scope for an 11/13-Fr or 10/12-Fr UAS. Stone fragmentation will be performed using a holmium laser (Ho: YAG) with a 272-μm fiber and an energy setting below 30 W. Irrigation will be maintained at 50-100 ml/min and suction pressure at 80-120 mmHg. at the end a 6 Fr JJ will be inserted for 4 weeks.
  Interventions: Procedure: Flexible Uerteroscopy with Tip-Bendable Suction Sheath

INTERVENTIONS:
Procedure: mini-percutaneous nephrolithotomy — Under general anesthesia, a 6 Fr ureteral catheter will be placed into the target ureter via cystoscopy, and bladder drainage will be achieved with a 16 Fr Foley catheter. The patient will then be repositioned to the prone position. Percutaneous renal access will be obtained by puncturing the selected calyx with an 18-gauge coaxial needle under fluoroscopic or ultrasound guidance. Tract dilation will be performed using fascial dilators up to 20 Fr then the mini-PCNL sheath (mini-Amplatz sheath) will be inserted and the mini nephroscope 12 to 15 Fr will be used. If multiple nephrostomy tracts are required for stone removal, the same approach will be repeated for each tract. Stone fragmentation will be carried out with a pneumatic lithotripter.
  At the end of the procedure, a 6 Fr double-J ureteral stent will be inserted for 4 weeks, and whether to place a nephrostomy tube will be determined at the discretion of the operating surgeon.
  Other Names: Mini-PCNL; mPCNL
  Arms: mini-PCNL
Procedure: Flexible Uerteroscopy with Tip-Bendable Suction Sheath — under general anesthesia with the patient in the lithotomy position. A 6 Fr ureteral catheter will first be placed into the ureter, followed by retrograde pyelography to assess the upper urinary tract. A guidewire will then be advanced into the renal pelvis. either a 12/14 Fr or 11/13 Fr tip-bendable S-UAS will be inserted. If insertion is not possible due to ureteral narrowing, a smaller 10/12 Fr UAS will be attempted. if failed, a double-J stent will be placed and the procedure terminated, with a second session scheduled 4 weeks later. fURS will be performed using digital flexible ureteroscopes either 8.5 Fr or 7.5 Fr according to UAS size; an 8.5-Fr scope for a 12/14 Fr UAS, and a 7.5-Fr scope for an 11/13-Fr or 10/12-Fr UAS. Stone fragmentation will be performed using a holmium laser (Ho: YAG) with a 272-μm fiber and an energy setting below 30 W. Irrigation will be maintained at 50-100 ml/min and suction pressure at 80-120 mmHg. at the end a 6 Fr JJ will be inserted for 4 weeks.
  Other Names: FANS; FURS with Suction Sheath
  Arms: FURS with Tip-Bendable Suction Sheath

SUMMARY:
This study aims to compare the efficacy and safety of two modern, minimally invasive surgical techniques for the removal of kidney stones: Mini-Percutaneous Nephrolithotomy (Mini-PCNL) and Flexible Ureteroscopy (FURS) with Flexible and navigable suction sheath

The primary objective is to determine which procedure results in a higher stone-free rate, as measured by post-operative imaging. Secondary objectives include comparing operative time, hospitalization length andcomplication rates between the two treatment groups.

Patients with two to three centimeter kidney stones who are candidates for either procedure will be randomly assigned to undergo either Mini-PCNL or suctioning FURS. The outcomes will be critically assessed to help establish a higher level of evidence for guiding surgical management of kidney stones.

DETAILED DESCRIPTION:
Mini-PCNL involves creating a small tract from the skin on the back directly into the kidney, through which a miniature nephroscope is passed to visualize and remove stones. Flexible Ureteroscopy is performed by passing a thin, flexible scope through the natural urinary passage (urethra and ureter) into the kidney. The specific FURS technique in this study utilizes a specialized scope with integrated suction, which is theorized to improve stone fragment clearance.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aging 18 years old or more.
* Patients with renal stones between 2-3 cm in size confirmed by CT scan.

Exclusion Criteria:

* Patients with previous ureteric injury.
* Patients with uncontrolled diabetes mellitus or hypertension.
* Patients with uncontrolled hepatic dysfunction.
* Patients with uremia or renal failure.
* Pregnant patients.
* patients with active urinary tract infection.
* Patients with bleeding tendency or uncontrolled coagulopathy.
* Patients with congenital anomalies as horse-shoe kidney and pelvi-ureteric junction obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
stone free rate | one month postoperative
  The proportion of participants in each treatment arm who are completely free of any stone fragments in the treated kidney, following the initial procedure and without the need for any secondary surgical interventions. Status will be determined by a blinded central radiologist.

SECONDARY OUTCOMES:
length of hospital stay | From date of surgery until date of hospital discharge for 14 days (measured in days).
  The total duration of inpatient hospitalization following the procedure, calculated from the day of surgery to the day of discharge
operative time | Measured intraoperatively, from procedure start to end (in minutes).
  The total time from the initiation of the procedure to the final removal of all endoscopic equipment and placement/completion of any necessary stents

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Tawfeek, assistant proffessor, Study Chair — Ain Shams University, Department Of Urology; Ahmed Higazy, lecturer of urology, Study Director — Ain Shams University, Department Of Urology; Ashraf Satour, lecturer of urology, Study Director — Ain Shams University, Department Of Urology
Locations (1):
- Ain shams university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhu W, Liu S, Cao J, Wang H, Liang H, Jiang K, Cui Y, Chai CA, Sahinler EB, Aquino A, Mazzon G, Zhong W, Zhao Z, Zhang L, Ding J, Wang Q, Wang Y, Chen KW, Liu Y, Choong S, Sarica K, Zeng G. Tip bendable suction ureteral access sheath versus traditional sheath in retrograde intrarenal stone surgery: an international multicentre, randomized, parallel group, superiority study. EClinicalMedicine. 2024 Jul 5;74:102724. doi: 10.1016/j.eclinm.2024.102724. eCollection 2024 Aug. PMID 39070176
- [Result] Tang QL, Liang P, Ding YF, Zhou XZ, Tao RZ. Comparative efficacy between retrograde intrarenal surgery with vacuum-assisted ureteral access sheath and minimally invasive percutaneous nephrolithotomy for 1-2 cm infectious upper ureteral stones: a prospective, randomized controlled study. Front Surg. 2023 Jul 7;10:1200717. doi: 10.3389/fsurg.2023.1200717. eCollection 2023. PMID 37483661
- [Result] Skolarikos A, Jung H, Neisius A, et al. EAU guidelines on urolithiasis. Arnhem, Netherlands: European Association of Urology; 2024.
- [Result] Pauchard F, Ventimiglia E, Corrales M, Traxer O. A Practical Guide for Intra-Renal Temperature and Pressure Management during Rirs: What Is the Evidence Telling Us. J Clin Med. 2022 Jun 15;11(12):3429. doi: 10.3390/jcm11123429. PMID 35743499
- [Result] Guven S, Yigit P, Tuncel A, Karabulut I, Sahin S, Kilic O, Balasar M, Seckiner I, Canda E, Sonmez MG, Tefik T, Boz MY, Atis G, Ergin G, Soytas M, Senel C, Kirac M, Kiremit MC, Akand M, Tugcu V, Erkurt B, Muslumanoglu A, Sarica K. Retrograde intrarenal surgery of renal stones: a critical multi-aspect evaluation of the outcomes by the Turkish Academy of Urology Prospective Study Group (ACUP Study). World J Urol. 2021 Feb;39(2):549-554. doi: 10.1007/s00345-020-03210-2. Epub 2020 Apr 28. PMID 32347334
- [Result] Geraghty R, Abourmarzouk O, Rai B, Biyani CS, Rukin NJ, Somani BK. Evidence for Ureterorenoscopy and Laser Fragmentation (URSL) for Large Renal Stones in the Modern Era. Curr Urol Rep. 2015 Aug;16(8):54. doi: 10.1007/s11934-015-0529-3. PMID 26077357
- [Result] Gauhar V, Traxer O, Castellani D, Sietz C, Chew BH, Fong KY, Hamri SB, Gokce MI, Gadzhiev N, Galosi AB, Yuen SKK, El Hajj A, Ko R, Zawadzki M, Sridharan V, Lakmichi MA, Corrales M, Malkhasyan V, Ragoori D, Soebhali B, Tan K, Chai CA, Tursunkulov AN, Tanidir Y, Persaud S, Elshazly M, Kamal W, Tefik T, Shrestha A, Tiong HC, Somani BK. Could Use of a Flexible and Navigable Suction Ureteral Access Sheath Be a Potential Game-changer in Retrograde Intrarenal Surgery? Outcomes at 30 Days from a Large, Prospective, Multicenter, Real-world Study by the European Association of Urology Urolithiasis Section. Eur Urol Focus. 2024 Dec;10(6):975-982. doi: 10.1016/j.euf.2024.05.010. Epub 2024 May 24. PMID 38789313
- [Result] Alenezi H, Denstedt JD. Flexible ureteroscopy: Technological advancements, current indications and outcomes in the treatment of urolithiasis. Asian J Urol. 2015 Jul;2(3):133-141. doi: 10.1016/j.ajur.2015.06.002. Epub 2015 Jun 23. PMID 29264133